CLINICAL TRIAL: NCT02795468
Title: The Usefulness of Ultrasound Guided Technique Insertion of Radial Artery Catheter in Neonates and Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jong Hwan Lee, Associate Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2016-03-128-001
Record Dates: First submitted 2016-05-26; First posted 2016-06-10 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Catheterization, Peripheral
Keywords: Peripheral; Arterial; Catheterization

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Palpation group (Active Comparator): The operator will use the pulsation of the radial artery as a guide for the cannulation.
  Interventions: Procedure: Radial arterial cannulation
- Ultrasound group (Experimental): The ultrasound guided technique will be used to find a radial artery and insert a radial arterial catheter.
  Interventions: Procedure: Radial arterial cannulation

INTERVENTIONS:
Procedure: Radial arterial cannulation — Radial arterial cannulation using usual palpation method or ultrasound guided technique according to the group

SUMMARY:
The investigators are trying to compare the ultrasound-guided technique vs. palpation method for radial arterial cannulation in infants.

DETAILED DESCRIPTION:
In infants (<12mo), radial arterial catheterization is sometimes difficult to perform. Moreover, repeated attempts itself would cause the arterial spasm or hematoma. The use of ultrasound as an adjunct to radial arterial cannulation has considered to be the best practice in adults and pediatrics. However, its usefulness or superiority for neonates and infants is not known. Therefore, we would compare ultrasound guided radial arterial cannulation with the usual palpation methods in infants undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Infants under 12 months age undergoing cardiac surgery with radial arterial cannulation

Exclusion Criteria:

* Sign of a skin infection
* Wound near the puncture site
* abnormal circulation of the hand
* any vascular problem at radial or ulnar artery

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2016-06; Primary Completion 2017-02 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
First-pass success rate | Within 10 min from the start time of arterial cannulation using an angiocath

CONTACTS AND LOCATIONS:
Overall Officials: Jong Hwan Lee, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Huang HP, Zhao WJ, Wen F, Li XY. Application of ultrasound-guided radial artery cannulation in paediatric patients: A systematic review and meta-analysis. Aust Crit Care. 2021 Jul;34(4):388-394. doi: 10.1016/j.aucc.2020.09.001. Epub 2020 Oct 21. PMID 33097369
- [Derived] Min JJ, Tay CK, Gil NS, Lee JH, Kim S, Kim CS, Yang JH, Jun TG. Ultrasound-guided vs. palpation-guided techniques for radial arterial catheterisation in infants: A randomised controlled trial. Eur J Anaesthesiol. 2019 Mar;36(3):200-205. doi: 10.1097/EJA.0000000000000926. PMID 30431501